CLINICAL TRIAL: NCT03103893
Title: Novel Compositions for Treating or Preventing Dermal Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1604004478
Record Dates: First submitted 2017-03-07; First posted 2017-04-06 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Dermal Atrophy
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Patients will apply lotions containing either rapamycin or vehicle to 2 distinct areas of sun exposed skin.
Masking Description: Clinical assessors are blinded to recruitment and treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rapamycin (Experimental): Rapamycin
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — topical formulation
  Other Names: sirolimus

SUMMARY:
This trial examines the impact of a topical formulation of rapamycin on dermal thickness and senescence.

DETAILED DESCRIPTION:
Aging of the skin is the most prominent feature of the aging process, being caused by multiple factors such as intrinsic aging process and UV light exposure.

Dermal atrophy, also called skin atrophy or atrophy, is a disorder manifesting thinning or depression of skin due to reduction of underlying tissue. Dermal atrophy is a major clinical problem in the elderly population. Loss of dermal integrity leads to increased fragility of the skin and precludes the use of intravenous lines in many cases. Skin tears are a significant concern in elderly individuals directly related to dermal atrophy. Impairment in wound healing is an important clinical sequelae of reduced dermal integrity leading to an increase in the number of the infections and complications following injury. Seborrheic keratosis, which comprise focal areas of epidermal thickening, can occur, possibly representing a response to damage. It has been estimated that 100% of individuals over 50 years of age harbor at least one of these lesion. There is not treatment for dermal atrophy and seborrheic keritoses require excision if they become large enough to cause discomfort or distress.

Therefore, there is a need to develop novel compositions and methods for treating or preventing certain age-related dermal conditions.

Rapamycin is an FDA approved drug that has been in clinical use for over 15 years. Systemic application of rapamycin has been a central part of immuno suppressive therapy for transplant patients in combination with other immuno suppressants. The safety record for systemic use of rapamycin is excellent and few side effects are associated with extended use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Individuals with any chronic disease will be excluded from the study including those with the following conditions:

  * Diabetes
  * Any type of Malignancy
  * Severe coronary artery disease
  * HIV infection
  * Hepatitis C or B
  * Any sign of skin disorder or disease aside from normal aging, dermal atrophy, or seborrheic keratoses.
  * Premenopausal women will be excluded
  * Patients taking the following medications will be excluded:
  * Cyclosporin
  * Calcium channel blockers: diltiazem, verapamil
  * Antifungal agents e.g. clotrimazole, fluconazole, itraconazole
  * Antibiotics: clarithromycin, erythromycin, rifampicin
  * Anticonvulsants: carbamazepine, phenobarbitone, phenytoin
  * Antinausea drugs e.g. metoclopramide
  * Other drugs e.g. danazol, protease inhibitors (e.g. for HIV and hepatitis C including ritonavir, indinavir, boceprevir, and telaprevir)
  * Grapefruit juice
  * St John's wort (Hypericum perforatum, hypericin)

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Dermal thickness | 6-8 months
  dermal thickness as assessed by direct measurement

SECONDARY OUTCOMES:
Gene expression | 6-8 months
  immunohistochemistry and gene expression analysis
Seborrheic Keratosis | 6-8 months
  clinical severity will be assess using a 1-5 rating scale of severity. Lesions will be evaluated for their progression over the treatment period relative to the known course of growth for Seborrheic Keratoses.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Sell, PhD, Principal Investigator — Faculty member; Christina Chung, MD, Principal Investigator — Drexel University College of Medicine; Ibiyonu Lawrence, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel Dermatology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung CL, Lawrence I, Hoffman M, Elgindi D, Nadhan K, Potnis M, Jin A, Sershon C, Binnebose R, Lorenzini A, Sell C. Topical rapamycin reduces markers of senescence and aging in human skin: an exploratory, prospective, randomized trial. Geroscience. 2019 Dec;41(6):861-869. doi: 10.1007/s11357-019-00113-y. Epub 2019 Nov 25. PMID 31761958